CLINICAL TRIAL: NCT07073131
Title: Comparison Between Maternal Complications of Chromic Catgut and Vicryl Rapid Sutures Used for Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huma Ijaz (Other)
Responsible Party: Sponsor-Investigator, Huma Ijaz, Dr Huma Ijaz, Combined Military Hospital Gujranwala
Organization: Combined Military Hospital Gujranwala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 37
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Episiotomy Extended by Laceration; Episiotomy Wound
Keywords: Episiotomy; Pain; Wound Infection
MeSH Terms: conditions — Pain; Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Vicryl Rapide suturing (Active Comparator): After approval from ethical review board (ERC letter no: 37-2024 dated 10-01-2024), 202 females fulfilling the selection criteria were enrolled from labor room. Informed consent was taken. Demographics were noted. Then participants underwent episiotomy. At end of procedure, they were randomly divided in two groups by using lottery method. Group A includes 101 participants that underwent suturing by using vicryl rapide. After 24 hours they were examined for pain score by using visual analogue scale. They were discharged after examining the episiotomy wound and were followed-up for 7 days in OPD. During follow-up, participants were examined for pain score, wound infection, inflammation and dehiscence.
  Interventions: Other: Vicryl Rapide suturing
- Participants with chromic catgut suturing (Active Comparator): Total 202 females fulfilling the selection criteria were enrolled from labor room. Informed consent was taken. Demographics were noted. Then participants underwent episiotomy. At end of procedure, they were randomly divided in two groups by using lottery method. Group B included 101 participants that underwent suturing by using chromic catgut. After 24 hours they were examined for pain score by using visual analogue scale. They were discharged after examining the episiotomy wound and were followed-up for 7 days in OPD. During follow-up, participants were examined for pain score, wound infection, inflammation and dehiscence.
  Interventions: Other: Chromic catgut suturing

INTERVENTIONS:
Other: Vicryl Rapide suturing — Post episiotomy vicryl rapide suturing material is used for stitching episiotomy laceration.
  Arms: Participants with Vicryl Rapide suturing
Other: Chromic catgut suturing — Post episiotomy chromic catgut suturing material is used for stitching episiotomy laceration
  Arms: Participants with chromic catgut suturing

SUMMARY:
Total 202 patients fulfilling the selection criteria were enrolled from labor room and underwent episiotomy. At end of procedure, females were randomly divided in two groups. In group A, females underwent suturing by using vicryl rapide. In group B, females underwent suturing by using chromic catgut. After 24 hours of delivery, females were examined for pain score. After 7 days, females were examined for wound infection, inflammation and dehiscence. All this information was recorded in proforma.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida of age 18-35 years
* Gestational age during 37-40 weeks

Exclusion Criteria:

* Females with abnormal placenta, non-cephalic presentation, multiple fetus, premature rupture of membranes, unclean vaginal examination.
* pre-delivery hemoglobin <9 g/dl,
* Manual removal of placenta
* Vulvar hematoma and vaginal tears

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 202 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Wound dehiscence | 7 days
  Wound dehiscence was labeled if there was partial or total separation of previously approximated wound edges, due to a failure of proper wound healing within 7 days of episiotomy.
Post surgical pain | 7 days
  After 24 hours of episiotomy participants were examined for pain score by using visual analogue scale.
Wound Infection | 7 days
  Wound infection was labeled if participant developed pain and pus discharge at wound site, along with fever (>100F) within 7 days of episiotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No